CLINICAL TRIAL: NCT02961751
Title: Clinical Validation of a Molecular Test for Ciprofloxacin-Susceptibility in Neisseria Gonorrhoeae
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 15-0090
Record Dates: First submitted 2016-11-09; First posted 2016-11-11 (Estimated); Results first posted 2020-01-29 (Actual); Last update posted 2020-08-25 (Actual); Status verified 2019-12-04

CONDITIONS: Gonococcal Infection
Keywords: Ciprofloxacin-susceptibility; Efficacy; Gyrase A Assay; Neisseria gonorrhoeae
MeSH Terms: conditions — Gonorrhea | interventions — Ciprofloxacin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Ciprofloxacin (Other): One dose of directly-observed ciprofloxacin 500 mg administered orally. N=381
  Interventions: Drug: Ciprofloxacin

INTERVENTIONS:
Drug: Ciprofloxacin — Directly observed treatment with a single dose of ciprofloxacin 500 mg orally with or without food.

SUMMARY:
This study is a multi-center, single-arm, open-label clinical study to assess the efficacy of one dose of ciprofloxacin given orally in subjects infected with untreated gyrase A (gyrA) serine 91 genotype Neisseria gonorrhoeae (N. gonorrhoeae) as determined by a real-time Polymerase Chain Reaction (PCR) assay. The study will enroll approximately 381 subjects to obtain an eligibility target of 257 subjects, per protocol, age 18 and older regardless of gender identification who are seeking care in Sexually Transmitted Disease (STD) clinics of up to eight of the participating sites in the United States. Subjects who have untreated gyrA serine 91 genotype N. gonorrhoeae of the rectum, or male or female urogenital tract identified by a positive culture or Nucleic Acid Amplification Test (NAAT) conducted at a prior visit will be offered enrollment in the study. They will receive one dose of directly observed ciprofloxacin 500 milligrams. Subjects not consenting to participate in the study will receive treatment per local standard of care. The duration of the study for each subject will be approximately 11 through 14 days. The primary objective of this study is to determine the efficacy of ciprofloxacin for treatment of uncomplicated N. gonorrhoeae infections with gyrA serine 91 genotype.

DETAILED DESCRIPTION:
This study is a multi-center, single-arm, open-label clinical study to assess the efficacy of one dose of ciprofloxacin given orally in subjects infected with untreated gyrase A (gyrA) serine 91 genotype Neisseria gonorrhoeae (N. gonorrhoeae) as determined by a real-time Polymerase Chain Reaction (PCR) assay. The study will enroll approximately 381 subjects to obtain an eligibility target of 257 subjects, per protocol, age 18 and older regardless of gender identification who are seeking care in Sexually Transmitted Disease (STD) clinics of up to eight of the participating sites in the United States. Subjects who have untreated gyrA serine 91 genotype N. gonorrhoeae of the rectum, or male or female urogenital tract identified by a positive culture or Nucleic Acid Amplification Test (NAAT) conducted at a prior visit will be offered enrollment in the study. They will receive one dose of directly observed ciprofloxacin 500 milligrams. Subjects not consenting to participate in the study will receive treatment per local standard of care. The duration of the study for each subject will be approximately 11 through 14 days. The primary objective of this study is to determine the efficacy of ciprofloxacin for treatment of uncomplicated N. gonorrhoeae infections with gyrA serine 91 genotype. The secondary objectives of the study are to 1) investigate the efficacy of ciprofloxacin for treatment of uncomplicated serine 91 gyrA N. gonorrhoeae infection by anatomic site and 2) to determine the sensitivity of the gyrA assay for detection of ciprofloxacin-susceptible N. gonorrhoeae infections.

ELIGIBILITY:
Inclusion Criteria:

1. Willing and able to give voluntary written informed consent before any study related procedure is performed.
2. 18 years or older, on the day of enrollment.
3. Untreated gyrA serine 91 genotype N. gonorrhoeae of the rectum, or male or female urogenital tract, as determined by the gyrA test assay on a specimen collected within 30 days of enrollment.

   *Subjects must have gyrA serine 91 genotype detected for N. gonorrhoeae from at least one non-pharyngeal site.
4. Willing to abstain from sexual intercourse or use condoms during any sexual contact until the Test of Cure Visit (Visit 2, Day 5-10) is complete.
5. Women of childbearing potential must have no vaginal intercourse 14 days before enrollment or use an effective birth control method for 30 days before enrollment and agree to continue through visit 2.

   *A woman is considered of childbearing potential unless post-menopausal (greater than 2 years) or surgically sterilized (tubal ligation greater than 1 year, bilateral oophorectomy, or hysterectomy).

   **Acceptable birth control methods for the purposes of this study may include abstinence from intercourse with a male partner, monogamous relationship with vasectomized partner, male condoms with the use of applied spermicide, intrauterine devices, and licensed hormonal methods. A highly effective method of contraception is defined as one that results in a low failure rate (i.e., less than 1 percent per year) when used consistently and correctly.
6. Able to swallow pills.
7. Willing to comply with protocol requirements, including availability for follow-up for the duration of the study.
8. Agree to avoid systemic or intravaginal antibiotics with activity against N. gonorrhoeae from enrollment through Visit 2 (Day 5-10). Topical and intravaginal antifungals are permitted.
9. Agree to avoid magnesium/aluminum antacids, sucralfate, didanosine, or highly buffered drugs, up to 2 hours after receipt of study drug.

Exclusion Criteria:

1. Known renal insufficiency from clinical history.
2. Use of systemic or intravaginal antibiotics with potential activity against N. gonorrhoeae within 30 days prior to study drug administration.

   *Topical and intravaginal antifungals are permitted.
3. Use of systemic corticosteroid drugs or other immunosuppressive therapy within 30 days prior to enrollment.
4. Receipt or planned receipt of an investigational product in a clinical trial within 30 days prior to or 7 days after treatment administration.
5. Pregnant or breastfeeding.
6. Clinical diagnosis of pelvic inflammatory disease or genital ulcer.
7. Confirmed or suspected complicated or systemic gonococcal infection, such as abdominal pain, testicular pain, epididymitis, orchitis, arthritis, or endocarditis.
8. Receipt of magnesium/aluminum antacids, sucralfate, didanosine, or highly buffered drugs, within 6 hours before receipt of study drug.
9. Mutant N. gonorrhoeae gyrA serine 91 genotype from any anatomic site, as determined by the gyrA test assay on a specimen collected within 30 days of enrollment.
10. Known allergy or history of adverse reaction to ciprofloxacin.
11. Known allergy to quinolones.
12. Previous enrollment in this study.
13. Medical condition or other factor that in the judgment of the investigator might affect ability to comply with procedures.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 211 (Actual)
Dates: Start 2016-10-19 (Actual); Primary Completion 2019-01-04 (Actual); Study Completion 2019-01-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (9):
- United States (9):
  - AIDS Healthcare Foundation Wellness Center - Hollywood, Los Angeles, California
  - Los Angeles Lesbian Gay Bisexual/Transgender Center, Los Angeles, California
  - University of California, San Diego - Antiviral Research Center, San Diego, California
  - University of California, San Diego Health - Owen Clinic, San Diego, California
  - San Francisco Department of Public Health - San Francisco City Clinic, San Francisco, California
  - Whitman-Walker Health, Washington D.C., District of Columbia
  - Louisiana State University Health Sciences Center, New Orleans, Louisiana
  - University of Mississippi - Infectious Diseases, Jackson, Mississippi
  - Philadelphia Department of Public Health - Health Center 1, Philadelphia, Pennsylvania

REFERENCES:
- [Derived] Klausner JD, Bristow CC, Soge OO, Shahkolahi A, Waymer T, Bolan RK, Philip SS, Asbel LE, Taylor SN, Mena LA, Goldstein DA, Powell JA, Wierzbicki MR, Morris SR. Resistance-Guided Treatment of Gonorrhea: A Prospective Clinical Study. Clin Infect Dis. 2021 Jul 15;73(2):298-303. doi: 10.1093/cid/ciaa596. PMID 32766725

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Sites/clinics recruited subjects from their existing patient population, patients that were sent by referral from other clinics, and walk-ins. 232 volunteers were screened to enroll 211 subjects between 13SEP2016 and 31DEC2018.
Groups:
- Ciprofloxacin: One dose of directly-observed ciprofloxacin 500 mg administered orally.
Period: Overall Study
Arm/Group | Ciprofloxacin
Started | 211
Completed | 196
Not Completed | 15
Not completed — Lost to Follow-up | 11
Not completed — Physician Decision | 2
Not completed — Not Eligible at Enrollment | 1
Not completed — Protocol Violation | 1

BASELINE CHARACTERISTICS:
Arm/Group | Ciprofloxacin
Number analyzed (Participants) | 211
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 211
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 28.9 (8.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21
  Male | 190
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 62
  Not Hispanic or Latino | 148
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 3
  Asian | 10
  Native Hawaiian or Other Pacific Islander | 2
  Black or African American | 70
  White | 103
  More than one race | 11
  Unknown or Not Reported | 12
Region of Enrollment [Number; unit: participants]
  United States | 211
Baseline Rectal/Urogenital Wild-Type N. gonorrhoeae infection [Count of Participants; unit: Participants] | 109
Baseline Urogenital Wild-Type N. gonorrhoeae infection [Count of Participants; unit: Participants] | 34
Baseline Rectal Wild-Type N. gonorrhoeae infection [Count of Participants; unit: Participants] | 79
Baseline Pharyngeal Wild-Type N. gonorrhoeae infection [Count of Participants; unit: Participants] | 16

OUTCOME MEASURES:

1. Primary Outcome: The Percentage of Subjects Infected With Gyrase A (gyrA) Serine 91 Genotype of Neisseria Gonorrhoeae (N. Gonorrhoeae) With Microbiological Cure
Description: Subjects infected with gyrase A (gyrA) serine 91 genotype of Neisseria gonorrhoeae (N. gonorrhoeae) were evaluated for microbiological cure at 5-10 days after treatment. Cure was defined as N. gonorrhoeae not detectable by culture from all anatomical sites that had detectable N. gonorrhoeae at baseline.
Time Frame: Day 5 through Day 10
Population: The per protocol population was limited to subjects meeting all inclusion criteria and no exclusion criteria and who were positive for rectal/urogenital wild type N. gonorrhoeae at baseline.
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | Ciprofloxacin
Number analyzed (Participants) | 99
percentage of subjects | 100 [97 to 100]

2. Secondary Outcome: The Percentage of Microbiologically Cured Subjects Who Had Urogenital Tract Infection Caused by gyrA Serine 91 Genotype N. Gonorrhoeae
Description: Subjects infected with gyrase A (gyrA) serine 91 genotype of Neisseria gonorrhoeae (N. gonorrhoeae) at the urogenital tract were evaluated for microbiological cure at 5-10 days after treatment. Cure was defined as N. gonorrhoeae not detectable by culture from all anatomical sites that had detectable N. gonorrhoeae at baseline
Time Frame: Day 5 through Day 10
Population: The per protocol population was limited to subjects meeting all inclusion criteria and no exclusion criteria and who were positive for urogenital wild type N. gonorrhoeae at baseline.
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | Ciprofloxacin
Number analyzed (Participants) | 30
percentage of subjects | 100 [90.5 to 100]

3. Secondary Outcome: The Percentage of Microbiologically Cured Subjects Who Had Rectal Infection Caused by gyrA Serine 91 Genotype N. Gonorrhoeae
Description: Subjects infected with gyrase A (gyrA) serine 91 genotype of Neisseria gonorrhoeae (N. gonorrhoeae) at the rectum were evaluated for microbiological cure at 5-10 days after treatment. Cure was defined as N. gonorrhoeae not detectable by culture from all anatomical sites that had detectable N. gonorrhoeae at baseline
Time Frame: Day 5 through Day 10
Population: The per protocol population was limited to subjects meeting all inclusion criteria and no exclusion criteria and who were positive for rectal wild type N. gonorrhoeae at baseline.
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | Ciprofloxacin
Number analyzed (Participants) | 73
percentage of subjects | 100 [96 to 100]

4. Secondary Outcome: The Percentage of Microbiologically Cured Subjects Who Had Throat Infection Caused by gyrA Serine 91 Genotype N. Gonorrhoeae
Description: Subjects infected with gyrase A (gyrA) serine 91 genotype of Neisseria gonorrhoeae (N. gonorrhoeae) at the throat were evaluated for microbiological cure at 5-10 days after treatment. Cure was defined as N. gonorrhoeae not detectable by culture from all anatomical sites that had detectable N. gonorrhoeae at baseline
Time Frame: Day 5 through Day 10
Population: The per protocol population was limited to subjects meeting all inclusion criteria and no exclusion criteria and who were positive for wild type N. gonorrhoeae of the throat at baseline.
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | Ciprofloxacin
Number analyzed (Participants) | 14
percentage of subjects | 100 [80.7 to 100]

5. Secondary Outcome: The Number of Subjects With Urethral Infection of gyrA Serine 91 Genotype N. Gonorrhoeae Who Have Ciprofloxacin-susceptible N. Gonorrhoeae
Description: Ciprofloxacin susceptibility was determined via culture-based antimicrobial susceptibility testing of the gonococcal isolate from each urethral sample with a positive N. gonorrhoeae culture at Visit 1. An infection was deemed susceptible to ciprofloxacin if the reported minimum inhibitory concentration for the isolate was < 1 mcg/ml. Detection of wild type gyrA was determined by the real-time PCR analysis of the gyrA gene from the swab taken at Visit 1.
Time Frame: Day 1
Population: Analysis population was intention-to-treat.
Measure: Count of Participants; unit: Participants
Arm/Group | Ciprofloxacin
Number analyzed (Participants) | 22
Participants | 22

6. Secondary Outcome: The Number of Subjects With Cervical Infection of gyrA Serine 91 Genotype N. Gonorrhoeae Who Have Ciprofloxacin-susceptible N. Gonorrhoeae
Description: Ciprofloxacin susceptibility was determined via culture-based antimicrobial susceptibility testing of the gonococcal isolate from each cervical sample with a positive N. gonorrhoeae culture at Visit 1. An infection was deemed susceptible to ciprofloxacin if the reported minimum inhibitory concentration for the isolate was < 1 mcg/ml. Detection of wild type gyrA was determined by the real-time PCR analysis of the gyrA gene from the swab taken at Visit 1.
Time Frame: Day 1
Population: Analysis population was intention-to-treat.
Measure: Count of Participants; unit: Participants
Arm/Group | Ciprofloxacin
Number analyzed (Participants) | 7
Participants | 7

7. Secondary Outcome: The Number of Subjects With Rectal Infection of gyrA Serine 91 Genotype N. Gonorrhoeae Who Have Ciprofloxacin-susceptible N. Gonorrhoeae
Description: Ciprofloxacin susceptibility was determined via culture-based antimicrobial susceptibility testing of the gonococcal isolate from each rectal sample with a positive N. gonorrhoeae culture at Visit 1. An infection was deemed susceptible to ciprofloxacin if the reported minimum inhibitory concentration for the isolate was < 1 mcg/ml. Detection of wild type gyrA was determined by the real-time PCR analysis of the gyrA gene from the swab taken at Visit 1.
Time Frame: Day 1
Population: Analysis population was intention-to-treat.
Measure: Count of Participants; unit: Participants
Arm/Group | Ciprofloxacin
Number analyzed (Participants) | 60
Participants | 60

8. Secondary Outcome: The Number of Subjects With Pharyngeal Infection of gyrA Serine 91 Genotype N. Gonorrhoeae Who Have Ciprofloxacin-susceptible N. Gonorrhoeae
Description: Ciprofloxacin susceptibility was determined via culture-based antimicrobial susceptibility testing of the gonococcal isolate from each pharyngeal sample with a positive N. gonorrhoeae culture at Visit 1. An infection was deemed susceptible to ciprofloxacin if the reported minimum inhibitory concentration for the isolate was < 1 mcg/ml. Detection of wild type gyrA was determined by the real-time PCR analysis of the gyrA gene from the swab taken at Visit 1.
Time Frame: Day 1
Population: Analysis population was intention-to-treat.
Measure: Count of Participants; unit: Participants
Arm/Group | Ciprofloxacin
Number analyzed (Participants) | 13
Participants | 13

ADVERSE EVENTS:
Time Frame: Adverse events were not collected for this study.
Description: Ciprofloxacin has a well-established safety profile and has been prescribed to several millions of people in the US and worldwide as it was the CDC's recommended treatment regimen for uncomplicated gonorrhea from 1993 to 2007. Therefore, adverse event assessment was not required for this study.
Arm/Group | Ciprofloxacin
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2018-12-17): https://cdn.clinicaltrials.gov/large-docs/51/NCT02961751/Prot_000.pdf
  • Statistical Analysis Plan (2019-04-08): https://cdn.clinicaltrials.gov/large-docs/51/NCT02961751/SAP_001.pdf